CLINICAL TRIAL: NCT02400827
Title: Study About Contamination of Ovarian Tissue by RT-PCR in Children With Solid Tumors.
Brief Title: Contamination of Ovarian Tissue by RT-PCR in Participants With Solid Tumors
Acronym: OVAMAR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: CHU-0229
Record Dates: First submitted 2015-03-24; First posted 2015-03-27 (Estimated); Last update posted 2015-03-27 (Estimated); Status verified 2015-03

CONDITIONS: Minimal Residual Disease; Fertility Preservation
Keywords: Polymerase Chain Reaction; fertility preservation
MeSH Terms: conditions — Neoplasm, Residual

GROUPS / COHORTS (1):
- cryopreservation
  Interventions: Other: malignant cells

INTERVENTIONS:
Other: malignant cells

SUMMARY:
For prepubertal patients, cryopreservation of ovarian tissue is the only option available to preserve their fertility before cancer treatment. But ovarian autograft raises the issue of the risk of reintroduction of potentially malignant cells. The aim of our study is to develop a specific and sensitive method for residual disease detection in the ovarian tissue from patients treated for a solid tumor during infancy, whose fertility may have been compromised by treatments and who benefited of ovarian tissue cryopreservation.

DETAILED DESCRIPTION:
Some solid tumors have high risk of metastatic localization including in ovaries. There is concern over the possible presence of malignant cells in ovarian tissue that could cause a recurrence of the primary disease after reimplantation. Thus, the possibility of ovarian tissue involvement needs to be evaluated with sensitive molecular methods. Those techniques are now available for leukaemia but histology is still the only way for solid tumors.

Based on our experience in detection by RT-PCR of minimal residual disease (MRD) in neuroblastoma since 1994 [Tchirkov et al. 2003] and in ovarian tissue cryopreservation since 1995 [Schubert et al. 2005, Chambon in press], we want to develop a specific and sensitive method for residual disease detection by RT-PCR in order to evaluate the tumor contamination of ovarian harvested tissue.

Study population: We chose 3 models of pediatric solid tumors with high risk of metastases and which often require sterilizing treatments (chemo and/or radiotherapy): neuroblastoma, Ewing tumor and alveolar rhabdosarcoma. We will use four tumor cells lines: IMR32 and SK-NSH for neuroblastoma; RD-ES for Ewing tumor; RH-30 for rhabdosarcoma. We plan to use 20 fragments per line.

Study duration: 12 months Study design: Ovarian tissue without known malignancy but with a condition warranting laparoscopy (benign cysts) will be harvested during kystectomy (perikystic tissue).

The harvested ovarian cortex will be cut: one half will be frozen according to our routine protocol [Schubert et al. 2005] and the other half will be contaminated with tumor cells lines. Then, detection of the specific transcript will be done by RT-PCR in fresh tissue and after freeze/thaw. Total RNA will be extracted with the TRI-reagent and qRT-PCR will be performed using the "TaqMan" technology.

Primary endpoint: to reach a sensitivity about 1/106 cells.

ELIGIBILITY:
Inclusion Criteria:

* Women of any age, diagnosed with a benign cyst that needs a laparoscopy may be included

Exclusion Criteria:

-

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: patients treated for a solid tumor during infancy
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2014-11; Primary Completion 2015-11 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
malignant cells about 1/10*6 cells. | at day 1

CONTACTS AND LOCATIONS:
Overall Officials: Justyna KANOLD, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France